CLINICAL TRIAL: NCT01947816
Title: HUMIRA® 40 mg Syringe 0.8 mL for Subcutaneous Injection Protocol for Special Investigation on Long-Term Administration Ulcerative Colitis
Brief Title: Special Investigation in Patients With Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P14-190
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2018-11

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Humira: Humira 40 mg (marketed product) eow for subcutaneous injection after initial dosage of 160 mg and 2nd dosage of 80 mg in two weeks after the initial administration, for up to 52 weeks.

SUMMARY:
This investigation will be conducted to obtain the following information regarding the use of Humira 40 mg Syringe 0.8 mL for Subcutaneous Injection in patients with Ulcerative Colitis.

1. Unknown adverse reactions (in particular, clinically significant)
2. Incidence and conditions of occurrence of adverse reactions in clinical practice
3. Factors likely to affect the safety and effectiveness

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving Humira for the first time for the treatment of Ulcerative Colitis

Exclusion Criteria:

Contraindications according to the Package Insert include patients who have any of the following:

* serious infections
* tuberculosis
* a history of hypersensitivity to any ingredient of Humira
* demyelinating disease or a history of demyelinating disease
* congestive cardiac failure

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients for the first time receiving Humira for the treatment of Ulcerative Colitis
Sampling Method: Non-Probability Sample
Enrollment: 1621 (Actual)
Dates: Start 2013-08-09 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1621 participants were enrolled. Among the enrolled participants, case report forms were not collected from 28 participants, and there were 1593 participants whose data in case report forms were assessable.
Groups:
- Humira: Humira 40 mg (marketed product) every other week (eow) for subcutaneous injection after initial dosage of 160 mg and 2nd dosage of 80 mg in two weeks after the initial administration, for up to 52 weeks.
Period: Overall Study
Arm/Group | Humira
Started (Number of participants with CRFs attained) | 1593
Completed (Number of participants not excluded from the safety and/or efficacy analysis sets) | 1523
Not Completed | 70

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Arm/Group | Humira
Number analyzed (Participants) | 1593
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 680
  Male | 913
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 1568
  Other Asians | 11
  Other (Not Specified) | 14
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/dL] — Population: participants with an assessment at the time of study drug administration start
  mg/dL
    number analyzed (Participants) | 1058
    (all) | 1.20 (2.35)
Mayo Score [Mean (Standard Deviation); unit: score on a scale] — The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment [PGA]), each of which ranges from 0 (normal) to 3 (severe disease). Population: participants with an assessment at the time of study drug administration start
  score on a scale
    number analyzed (Participants) | 168
    (all) | 7.5 (2.3)
Endoscopy Results [Count of Participants; unit: Participants] — The endoscopist evaluated each observed segment of the colon (rectum, sigmoid, descending colon, transverse colon, ascending colon/cecum) by using the classification as follows: 0=Normal or inactive disease; 1=Mild disease (erythema, decreased vascular pattern, mild friability); 2=Moderate disease (marked erythema, absent vascular pattern, friability, erosions); 3=Severe disease (spontaneous bleeding, ulceration). Population: participants with an assessment at the time of study drug administration start
  Participants
    Normal or Remission-Phase Mucosa: number analyzed (Participants) | 179
    Normal or Remission-Phase Mucosa | 3
    Mild: number analyzed (Participants) | 179
    Mild | 11
    Moderate: number analyzed (Participants) | 179
    Moderate | 104
    Severe: number analyzed (Participants) | 179
    Severe | 61
Partial Mayo Score [Mean (Standard Deviation); unit: score on a scale] — The Partial Mayo score (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment [PGA]), each of which ranges from 0 (normal) to 3 (severe disease). Population: participants with an assessment at the time of study drug administration start
  score on a scale
    number analyzed (Participants) | 1186
    (all) | 5.1 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions and Serious Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events for which the causal relation with Humira cannot be ruled out. Serious adverse drug reactions are adverse drug reaction(s) which have been assessed to be serious based on company criteria.
Time Frame: Up to Week 52
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Humira
Number analyzed (Participants) | 1523
Participants
  Adverse Drug Reactions | 276
  Serious Adverse Drug Reactions | 74

2. Secondary Outcome: Change From Baseline in CRP Levels Over Time
Time Frame: Weeks 4, 8, 24, 52 of study drug administration, and at study drug discontinuation (up to Week 52)
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Humira
Number analyzed (Participants) | 882
mg/dL
  Week 4 | 0.64 (1.65)
  Week 8: number analyzed (Participants) | 773
  Week 8 | 0.53 (1.34)
  Week 24: number analyzed (Participants) | 533
  Week 24 | 0.38 (1.00)
  Week 52: number analyzed (Participants) | 597
  Week 52 | 0.29 (0.89)
  At Discontinuation: number analyzed (Participants) | 308
  At Discontinuation | 2.10 (3.68)

3. Secondary Outcome: Change From Baseline in Mayo Score Over Time
Description: The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment [PGA]), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Weeks 24, 52, at study drug discontinuation (up to Week 52), and at final assessment (up to Week 52)
Population: participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Humira
Number analyzed (Participants) | 168
score on a scale
  Week 24: number analyzed (Participants) | 56
  Week 24 | -4.4 (3.1)
  Week 52: number analyzed (Participants) | 99
  Week 52 | -4.8 (3.1)
  When Discontinued: number analyzed (Participants) | 41
  When Discontinued | 0.8 (3.5)
  At Final Assessment | -3.3 (4.0)
Statistical Analysis 1: Comparison: Humira; Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, paired t-test
Statistical Analysis 2: Comparison: Humira; Change from Baseline at Week 52; Test type: Superiority; p < 0.0001, paired t-test
Statistical Analysis 3: Comparison: Humira; Change from Baseline When Discontinued; Test type: Superiority; p = 0.5512, paired t-test
Statistical Analysis 4: Comparison: Humira; Change from Baseline at Final Assessment; Test type: Superiority; p < 0.0001, paired t-test

4. Secondary Outcome: Mayo Endoscopic Sub-Score Over Time
Description: The endoscopist evaluated each observed segment of the colon (rectum, sigmoid, descending colon, transverse colon, ascending colon/cecum) by using the classification as follows: 0=Normal or inactive disease; 1=Mild disease (erythema, decreased vascular pattern, mild friability); 2=Moderate disease (marked erythema, absent vascular pattern, friability, erosions); 3=Severe disease (spontaneous bleeding, ulceration).
Time Frame: Weeks 24, 52, at study drug discontinuation (up to Week 52), and at final assessment (up to Week 52)
Population: participants with an assessment at given time point
Measure: Count of Participants; unit: Participants
Arm/Group | Humira
Number analyzed (Participants) | 179
Participants
  Week 24: number analyzed (Participants) | 61
  Week 24: 0=Normal or Inactive Disease | 18
  Week 24: 1=Mild Disease | 21
  Week 24: 2=Moderate Disease | 16
  Week 24: 3=Severe Disease | 6
  Week 52: number analyzed (Participants) | 102
  Week 52: 0=Normal or Inactive Disease | 35
  Week 52: 1=Mild Disease | 34
  Week 52: 2=Moderate Disease | 29
  Week 52: 3=Severe Disease | 4
  When Discontinued: number analyzed (Participants) | 46
  When Discontinued: 0=Normal or Inactive Disease | 2
  When Discontinued: 1=Mild Disease | 5
  When Discontinued: 2=Moderate Disease | 21
  When Discontinued: 3=Severe Disease | 18
  At Final Assessment: 0=Normal or Inactive Disease | 47
  At Final Assessment: 1=Mild Disease | 49
  At Final Assessment: 2=Moderate Disease | 58
  At Final Assessment: 3=Severe Disease | 25

5. Secondary Outcome: Change From Baseline in Partial Mayo Score Over Time
Description: The Partial Mayo score (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment [PGA]), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Partial Mayo score indicates improvement.
Time Frame: Weeks 4, 8, 16, 24, 52, when discontinued (up to Week 52), at final assessment (up to Week 52)
Population: participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Humira
Number analyzed (Participants) | 1186
score on a scale
  Week 4: number analyzed (Participants) | 1068
  Week 4 | -2.1 (2.4)
  Week 8: number analyzed (Participants) | 935
  Week 8 | -2.5 (2.6)
  Week 16: number analyzed (Participants) | 765
  Week 16 | -2.8 (2.6)
  Week 24: number analyzed (Participants) | 697
  Week 24 | -3.0 (2.6)
  Week 52: number analyzed (Participants) | 724
  Week 52 | -3.5 (2.6)
  When Discontinued: number analyzed (Participants) | 376
  When Discontinued | -0.7 (2.7)
  At Final Assessment | -2.5 (3.0)
Statistical Analysis 1: Comparison: Humira; Change from Baseline at Week 4; Test type: Superiority; p < 0.0001, paired t-test
Statistical Analysis 2: Comparison: Humira; Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, paired t-test
Statistical Analysis 3: Comparison: Humira; Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, paired t-test
Statistical Analysis 4: Comparison: Humira; Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, paired t-test
Statistical Analysis 5: Comparison: Humira; Change from Baseline at Week 52; Test type: Superiority; p < 0.0001, paired t-test
Statistical Analysis 6: Comparison: Humira; Change from Baseline when discontinued; Test type: Superiority; p < 0.0001, paired t-test
Statistical Analysis 7: Comparison: Humira; Change from Baseline at Final Assessment; Test type: Superiority; p < 0.0001, paired t-test

ADVERSE EVENTS:
Time Frame: up to Week 52
Arm/Group | Humira
All-Cause Mortality (participants affected / at risk) | 5/1523
Serious Adverse Events (participants affected / at risk) | 74/1523
Other Adverse Events (participants affected / at risk) | 0/1523
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Humira (N=1523)
Cellulitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2)
Cytomegaloviral infections (Infections and infestations) | 1 (1)
Disseminated tuberculosis (Infections and infestations) | 1 (1)
Endotoxic shock (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Gastroenteritis staphylococcal (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Liver abscess (Infections and infestations) | 2 (2)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonia influenzal (Infections and infestations) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 1 (1)
Cytomegalovirus enterocolitis (Infections and infestations) | 2 (2)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Infective thrombosis (Infections and infestations) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Infective spondylitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Cytomegalovirus mucocutaneous ulcer (Infections and infestations) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 (2)
Aspergillus infection (Infections and infestations) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Granulocytopenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Dermatopathic lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 2 (2)
Takayasu's arteritis (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 18 (18)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 2 (2)
Megacolon (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 5 (5)
Renal haemorrhage (Renal and urinary disorders) | 1 (1)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 2 (2)
Pyrexia (General disorders) | 5 (5)
C-reactive protein increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
C-reactive protein abnormal (Investigations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT01947816/SAP_000.pdf
  • Study Protocol (2018-04-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT01947816/Prot_001.pdf